CLINICAL TRIAL: NCT05774353
Title: Patients' Choice of Health Care Provider for Monitoring Their Pregnancy
Acronym: Grossesse-Cx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRD0322
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Pregnancy monitoring; Healthcare professional
MeSH Terms: interventions — Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient questionnaire (Other): Patients included in the study will complete an online questionnaire (LimeSurvey).
  Interventions: Other: Patient questionnaire

INTERVENTIONS:
Other: Patient questionnaire — Patients included in the study will complete an online questionnaire (LimeSurvey).

SUMMARY:
The aim of this study is to understand and interpret the determinants that lead pregnant women to refer more to a health professional in order to better meet the patient's request.

DETAILED DESCRIPTION:
Pregnancy is a natural phenomenon that occurs without complication in the majority of pregnant women. Pregnancy monitoring is necessary to detect possible complications and improve the comfort and experience of all pregnant women. For several years now, pregnant women have wanted to benefit from pregnancy monitoring as well as a less medical and physiological delivery according to the perinatal plan 2005-2007.

Perinatal plans have been implemented and evaluated for over 30 years. Progress has been made in terms of obstetrical and perinatal safety. The latest plan advocates a "humanisation of birth" which leaves more room for the parents' wishes. Pregnancy monitoring is currently carried out by doctors or midwives as part of seven compulsory prenatal examinations. This medical follow-up is completed by a preparation for birth with group classes, based on these general and obstetrical assessments.

After declaring their pregnancy, women can consult various health professionals to monitor their pregnancy. The aim of this study is to understand and interpret the determinants that lead pregnant women to be more oriented towards one health professional or another. Each determinant will be analysed and quantified in order to better respond to patient demand. The investigator chose to interview women who had just given birth and not pregnant women because the health professional may change during the course of the pregnancy, and the investigator assumes that the women will have more perspective on their experience and their choice once they have given birth.

ELIGIBILITY:
Inclusion Criteria :

* Woman in post-natal care at the NOVO hospital - Pontoise site
* Women aged 18 and over

Exclusion Criteria :

* Women who do not speak or understand French language (written and oral)
* Woman under legal protection (guardianship, curatorship...)
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is aimed at women who have just given birth at the NOVO hospital - Pontoise site
Enrollment: 400 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Determine which healthcare professional would be preferred by women who have just given birth, for the follow-up of their next possible pregnancy. | At the end of the study, an average of 6 month
  The healthcare professional preferred by the patients for the monitoring of their next pregnancy will be determined by the online questionnaire: question number 20.
  Question 20 : In the event of a future pregnancy, which health professional would you like to be followed by? Choice of answer : Medical gynaecologist, Obstetric gynaecologist, General practitioner and Midwife.

SECONDARY OUTCOMES:
Assessment of the influence of the presence or absence of risk factors on the choice of healthcare professional | At the end of the study, an average of 6 month
  The presence or absence of risk factors (hypertension, obesity, history of premature birth, history of caesarean section, etc.) will be sought in the patient's medical file
Assessment of the influence of the acquaintance of the healthcare professional before pregnancy monitoring on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the acquaintance of the healthcare professional on the choice of the healthcare professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 11.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the acquaintance of the healthcare professional before pregnancy monitoring". Choice of answer : Not important, Not very important, Important, Very important.
  Question 11: For how many years have you known the professional who has followed you the most during your pregnancy? Choice of answer : less than 5 years, between 5 and 10 years or more than 10 years.
Assessment of the influence of the gender of the healthcare professional on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the gender of the health professional on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 12.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the gender of the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 12: Do you have a preference regarding the gender of the health professional? If so, which one? Choice of answer : No preference, Male or Femal.
Assessment of the influence of the age of the healthcare professional on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the age of the health professional on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 13.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the age of the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 13: In your opinion, the ideal age of the health professional who follows your pregnancy is? Choice of answer : less than 40 years, between 40 and 60 years, more than 60 years or no preference.
Assessment of the influence of the availability of the healthcare professional on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the availability (particularly delay to make an appointment) of the health professional on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 14.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the availability of the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 14: Apart from the monthly follow-up, an appointment time with the health professional is appropriate if it is? Choice of answer : within 48 hours, within 7 days or within 15 days.
Assessment of the influence of the reachability of the healthcare on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the reachability of the health professional on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 15.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the reachability of the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 15: In choosing your health professional, a waiting period for advice is appropriate if it is? Choice of answer : within 24 hours, within 48 hours or within 7 days.
Assessment of the influence of the distance from physician's office to home (or work) on the choice of healthcare professional | At the end of the study, an average of 6 month
  distance from physician's office to home (or work) on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 16.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the distance from physician's office to home (or work)". Choice of answer : Not important, Not very important, Important, Very important.
  Question 16: In choosing your health professional, the distance from physician's office to home (or work) is appropriate if it is? Choice of answer : less than 15 minutes, between 15 and 29 minutes, between 30 and 44 minutes or more than 45 minutes.
Assessment of the influence of the price of the consultation of the healthcare professional on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the price of the consultation on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 17.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the price of the consultation of the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 17: In choosing your health professional, the price of the consultation is appropriate if it is? Choice of answer : less than 29 euros, between 30 and 59 euros, between 60 and 89 euros or 90 euros and more.
Assessment of the influence of time spent with the healthcare professional on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the of time spent with the healthcare professional on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 18.
  Question 10: In choosing your health care provider for your pregnancy follow-up, what are the important determinants and characteristics in your opinion? For "the time spent with the healthcare professional". Choice of answer : Not important, Not very important, Important, Very important.
  Question 18: In choosing your health professional, the time spent with the healthcare professional is appropriate if it is? Choice of answer : less than 15 minutes, between 15 and 29 minutes, between 30 and 44 minutes or 45 minutes and more.
Assessment of the influence of the healthcare professional's skills on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the healthcare professional's skills on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 10 and 19.
  Question 10: For "the healthcare professional's skills". Choice of answer : Not important, Not very important, Important, Very important.
  Question 19: Prioritise the most important competences of the health professional: (between 1 and 9, number 1 being the most important skill) Choice of skill : Caring attitude, empathy (does he put himself in your shoes?), Adapted and accessible communication (simple, understandable words), Diplomas/training, reliable information (without errors), Listening to the patient's wishes (shared decisions), Easily reachable professional, Patience, Pedagogy (explanations), Punctualitý and Decision-making
Assessment of the influence of the ultrasound practice in the physician's office on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of ultrasound practice in the physician's office on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: question number 10.
  Question 10: For "the ultrasound practice in the physician's office". Choice of answer : Not important, Not very important, Important, Very important.
Assessment of the influence of the possibility of following the child after birth on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the possibility of following the child after birth on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: question number 10.
  Question 10: For "the possibility of following the child after birth". Choice of answer : Not important, Not very important, Important, Very important.
Assessment of the influence of the setting of the physician's office on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the setting of the physician's office (equipment, size of the office, Secretariat) on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: question number 10.
  Question 10: For "the setting of the physician's office". Choice of answer : Not important, Not very important, Important, Very important.
Assessment of the influence of the follow-up with the attending physician on the choice of healthcare professional | At the end of the study, an average of 6 month
  The evaluation of the influence of the follow-up with the attending physician on the choice of the health professional for the monitoring of their next pregnancy will be determined by the online questionnaire: questions number 21 to 28.
  Q21: Do you have a follow-up with a general practitioner outside of pregnancy? Q22 :How old is your general practitioner? Q23 : How many years have you known him/her? Q24 :How do you feel about being treated by your general practitioner outside of pregnancy? Q25 : Does he/she practice gynaecology (screening, cervico-uterine smears, contraception...)? Q26 :Has he/she ever offered to monitor your pregnancy? Q27 :Do you think he/she is sufficiently trained in pregnancy monitoring? Q28 : In your opinion, is it the role of the general practitioner to provide gynaecological follow-up during and outside pregnancy?

CONTACTS AND LOCATIONS:
Overall Officials: Pr Christophe Poncelet, Principal Investigator — Hospital NOVO - Pontoise site
Locations (1):
- Gynaecology and obstetrics department - Hospital NOVO - Pontoise site, Pontoise, France

REFERENCES:
- See also: 4. Haut Conseil de la Santé Publique, ADSP (Actualité et dossier en santé publique) n° 61/62, Naître en France, 2007 — https://www.hcsp.fr/explore.cgi/adsp?clef=102
- See also: Le plan de périnatalité 2005-2007 : humanité, proximité, sécurité, qualité — http://portail.naissance.asso.fr/docs/planperinat.pdf
- See also: Service Public, Grossesse : examens médicaux, 2022 — https://www.service-public.fr/particuliers/vosdroits/F963
- See also: La moitié des rendez-vous sont obtenus en 2 jours chez le généraliste, en 52 jours chez l'ophtalmologiste — https://drees.solidarites-sante.gouv.fr/publications/etudes-et-resultats/la-moitie-des-rendez-vous-sont-obtenus-en-2-jours-chez-le
- See also: Recommandation HAS, Comment mieux informer les femmes enceintes — https://www.has-sante.fr/jcms/c_454394/fr/comment-mieux-informer-les-femmes-enceintes